CLINICAL TRIAL: NCT05889949
Title: Prediction of Microvascular Invasion by Radiomics Based on Pre-treatment Magnetic Resonance Imaging (MRI) for Guiding Treatment of Barcelona Clinic Liver Cancer (BCLC) Stage B Hepatocellular Carcinoma (HCC): A Prospective Cohort Study
Brief Title: Microvascular Invasion for Guiding Treatment of Barcelona Clinic Liver Cancer Stage B Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Professor, Sun Yat-sen University
Other Study IDs: HCC 007
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Radiomics; Hepatocellular Carcinoma (HCC); Transcatheter Arterial Chemoembolization (TACE); Microvascular Invasion (MVI); Multi-kinase Inhibitors (MKI)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE+MKIs
  Interventions: Drug: Sorafenib; Drug: Lenvatinib
- TACE

INTERVENTIONS:
Drug: Sorafenib — oral sorafenib
  Groups: TACE+MKIs
Drug: Lenvatinib — oral lenvatinib
  Groups: TACE+MKIs

SUMMARY:
The goal of this observational study is to explore the role of prediction of microvascular invasion by radiomics based on pre-treatment magnetic resonance imaging for guiding treatment of Barcelona Clinic Liver Cancer stage B hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. BCLC stage B HCC;
3. Received no previous anti-cancer treatment;
4. At least 1 measurable intrahepatic lesion based on the Response Evaluation Criteria in Solid Tumors criteria (RECIST) 1.1;
5. Adequate hematological, liver, renal function:

   1. absolute neutrophil count ≥ 1.5×109/L;
   2. platelet count ≥ 100×109/L;
   3. hemoglobin concentration ≥ 90 g/L;
   4. albumin ≥ 28 g/L;
   5. total bilirubin < 1.5 times the upper limit of normal;
   6. alanine aminotransferase and aspartate aminotransferase < 5 times the upper limit of normal;
   7. blood urea nitrogen and serum creatinine concentration < 1.5 times the upper limit of the normal range or less and creatinine clearance rate ≥ 45 mL/min;
6. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Acute or chronic active hepatitis B (HBV) or C (HCV) infection with HBV-DNA > 2000 IU/ml or 104 copies/ml; hepatitis C virus RNA > 103 copies/ml; HBsAg and anti-HCV antibody positive at the same time. Those who are below the above criteria after nucleoside based antiviral therapy may be enrolled;
2. Life-threatening bleeding event within the past 3 months, including the need for blood transfusion, surgical or local treatment, or continuous medication;
3. History of previous arterial or venous thromboembolic events within the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary artery embolism, deep vein thrombosis, or any other serious thromboembolism;
4. Use of aspirin (>325 mg/day) or other drugs known to inhibit platelet function such as dipyridamole or clopidogrel for 10 consecutive days within 2 weeks prior to enrollment;
5. Uncontrolled hypertension, systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy;
6. Symptomatic congestive heart failure (New York Heart Association class II-IV); Symptomatic or poorly controlled arrhythmias; History of congenital long QT syndrome or corrected QT (QTc) > 500 ms at screening;
7. Diagnosis of other malignant tumors within 5 years prior to enrollment;
8. Pregnant or lactating women or subjects planning to have a baby during the study period;
9. Accompanied with other uncontrolled co-morbidities;
10. Co-infection with HIV, known syphilis infection requiring treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BCLC stage B HCC patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of enrollment to the date of death due to any cause or last follow-up, whichever came first, assessed up to 48 months
  OS was defined as the interval from the date of enrollment to the date of death due to any cause or last follow-up.
Progression-Free Survival (PFS) | From the date of enrollment to the date of disease progression or the date of death due to any cause or last follow-up, whichever came first, assessed up to 48 months
  PFS was defined as the interval from the date of enrollment to the date of disease progression or the date of death due to any cause or last follow-up, whichever occurred first.

SECONDARY OUTCOMES:
Tumor response | From the date of enrollment to the date of death due to any cause or last follow-up, whichever came first, assessed up to 48 months
  Assessed by enhanced CT or MR at baseline, every 6 weeks after treatment initiation, using RECIST 1.1 The assessment of tumor response was performed independently by two experienced radiologists who were blinded to the patient's clinical information, and any inconsistent assessment results were resolved by further consensus.
Adverse events | From the date of enrollment to the date of death due to any cause or last follow-up, whichever came first, assessed up to 48 months
  The severity of adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE v5.0) .

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China